CLINICAL TRIAL: NCT02196051
Title: Lipid and Carbohydrate Metabolism: Effects of Exercise
Brief Title: Basic Research Study to Examine the Relation Between Muscle Insulin Resistance and Lipid Production in the Liver.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0710003207; R56AG023686 (NIH)
Record Dates: First submitted 2014-06-25; First posted 2014-07-21 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Insulin Resistance
Keywords: Insulin resistance; Exercise; de novo lipogenesis; NAFLD; Magnetic Resonance Spectroscopy
MeSH Terms: conditions — Insulin Resistance; Motor Activity; Non-alcoholic Fatty Liver Disease | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Training (Experimental): Participants engaged in a single bout of elliptical exercise for 45 minutes (3 times 15 minutes spaced by 5 minutes rest) at baseline. Subjects will be studied before and after this one bout to measure hepatic de novo lipogenesis. Hepatic de novo lipogenesis will be compared pre and post to examine whether acutely improving muscle glucose uptake will decrease hepatic de novo lipogenesis as the glucose is taken up by muscle and not directed to the liver.
  Interventions: Other: one bout of 45 minutes exercise

INTERVENTIONS:
Other: one bout of 45 minutes exercise — 45 minutes of exercise on an elliptical exercise machine

SUMMARY:
The purpose of this study was to examine the pathophysiology of insulin resistance and the relation to the metabolic syndrome in humans.

DETAILED DESCRIPTION:
In this study insulin resistant (IR), young offspring of parents with type 2 diabetes (18-46 years) and healthy, lean elderly individuals (65-90 years) underwent 1H/13C MRS measurements of liver and muscle lipid and glycogen content before and after a high carbohydrate meal challenge. Hepatic de novo lipogenesis was determined as the incorporation of deuterium, from deuterium labeled water (2H2O), into plasma triglycerides 5. These metabolic studies were performed in 2 sets: Study Part 1: Resting, Study Part 2: After 1 bout of 45 minutes exercise.

The study has been completed and published as two papers: August 16, 2011 and July 24, 2012.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index < 29 kg/m2
* No regular exercise routine
* Non-smokers
* Absence of systemic and organ disease.

Exclusion Criteria:

* Hematocrit < 35 vol%
* History of claustrophobia
* Ferromagnetic implants
* Regular exercise regimen
* Not weight stable
* Any significant hematological, neurological, musculoskeletal or endocrine disease (including diabetes mellitus)
* Any significant cardiovascular condition, including confirmed CAD and prior cardiovascular events
* Taking coumadin as anticoagulant therapy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2012-01-30 (Actual); Study Completion 2012-01-30 (Actual)

PRIMARY OUTCOMES:
change in de novo lipogenesis | Baseline
  At the baseline assessment, de novo lipogenesis was assessed after a high carbohydrate meal and a drink of heavy water. Muscle glycogen and lipid contents were measured pre- and post meal using 1H/13C MRS and de novo lipogenesis was assessed from the heavy water incorporation into blood lipid in samples collected overnight.

CONTACTS AND LOCATIONS:
Overall Officials: Kitt Petersen, MD, Principal Investigator — Yale University
Locations (1):
- YCCI/YNNH Hospital Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rabol R, Petersen KF, Dufour S, Flannery C, Shulman GI. Reversal of muscle insulin resistance with exercise reduces postprandial hepatic de novo lipogenesis in insulin resistant individuals. Proc Natl Acad Sci U S A. 2011 Aug 16;108(33):13705-9. doi: 10.1073/pnas.1110105108. Epub 2011 Aug 1. PMID 21808028
- [Result] Flannery C, Dufour S, Rabol R, Shulman GI, Petersen KF. Skeletal muscle insulin resistance promotes increased hepatic de novo lipogenesis, hyperlipidemia, and hepatic steatosis in the elderly. Diabetes. 2012 Nov;61(11):2711-7. doi: 10.2337/db12-0206. Epub 2012 Jul 24. PMID 22829450